CLINICAL TRIAL: NCT03285789
Title: Evaluation of the Visuo-attention Field of Symbols Versus Objects Visual Search in Dyslexic Subjects. DyslexiaSPOTLIGHT
Brief Title: Dyslexics' Visual Attention Field
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0333; 2017-A02525-48 (Other: ID-RCB)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Dyslexia
Keywords: Dyslexia; Visual Fields; visual attention span; visual search; visual attention field
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dyslexics with reduced visual attention span (Experimental): 21 subjects diagnosed dyslexics with reduced visual attention span
  Interventions: Other: Passing tests in dyslexics with reduced eva
- Dyslexics with normal visual attention span (Experimental)
  Interventions: Other: Passing tests in dyslexics with reduced eva
- controls (Active Comparator)
  Interventions: Other: Passing tests in controls

INTERVENTIONS:
Other: Passing tests in dyslexics with reduced eva — Visual attention span : the subject see a 5 letters strings during 200 ms and he has to report it orally whatever the order Visual search : the subject has to find a target among distractors (24 or 48) in different conditions of stimuli (conjunction feature or separable feature) and different conditions of view (full view or reduced view with the moving window paradigm) Elementary visuo spatial perception: the subject passes 6 visuo spatial tests to judge his visuo spatial abilities.
  All of these tests will be made during an unique visit of 1h30.
  Arms: Dyslexics with normal visual attention span; Dyslexics with reduced visual attention span
Other: Passing tests in controls — Visual attention span : the subject see a 5 letters strings during 200 ms and he has to report it verbally whatever the order Visual search : the subject has to find a target among distractors (24 or 48) in different conditions of stimuli (conjunction feature or separable feature) and different conditions of view (full view or reduced view with the moving window paradigm) Elementary visuo spatial perception: the subject passes 6 visuo spatial test to judge his visuo spatial abilities.
  "test de l'alouette" : reading test during 3 minutes, we note the number of word read and the errors. We obtain lexical age.
  All of these tests will be made during an unique visit of 1h30.
  Arms: controls

SUMMARY:
dyslexia is often considered like a phonological deficit but some researches show that a visual attention (V-A) deficit can occur in dyslexia. The investigator want to show that some dyslexics have a reduced V-A field in visual search when the investigator use separable feature (letter-like).

If the investigator demonstrate that, he will show that V-A deficit can be transpose to an ability acquired before reading, the visual search. Therefore, the V-A deficit can't be a consequence of reading problem but a cause of it for some dyslexics.

The investigator could imagine an earlier diagnosis for children at risk to develop dyslexia and make reeducation more specific for the deficit observed.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal vision
* diagnosed dyslexics with a recent "alouette" test

Exclusion Criteria:

* other developmental problem (dysphasia, dyspraxia, ADHD)
* strabismus, amblyopia, oculomotor paralysis

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1460 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Respond time in visual search in different condition of view (full view or reduced view) with separable feature. | Day 0
  The subject will have to find a target among distractors, when he will find it, he will have to push a button and we will have his respond time. We will compare the respond time in two view condition: the participant will see all the visual scene or he will have reduced visible window so he won't see all the scene, the periphery will be hide and he will have to move his sight to show it.

SECONDARY OUTCOMES:
respond time in function of the distractors' number | Day 0
  The subject will have to find a target among distractors, when he will find it, he will have to push a button and we will collect his respond time. We compare the respond time between two number of distractors (24 or 48)
visual exploration of the scene | Day 0
  with an eye tracker the investigator will analyze the ocular movements during visual search (saccades and fixations) and the equip will compare the visual behavior between the different groups and the different conditions.
visuo-spatial perception | Day 0
  the investigator will test with different exercises the elementary visuo spatial perception of the participant and he will compare between groups and also he will make correlation with the respond time in visual search.
visual attention span (VAS) | Day 0
  the subject have to report orally a 5 letters' string presented during 200 ms, the investigator could see if a correlation exist between VAS and RT, VAS and visual exploration, VAS and visuo spatial perception.

CONTACTS AND LOCATIONS:
Overall Officials: Laure PISELLA, PhD, Principal Investigator — INSERM U1028 - Impact - CRNL
Locations (1):
- U1028 INSERM - CNRS UMR 5292 Equipe ImpAct, Bron, France